CLINICAL TRIAL: NCT00005709
Title: Lipoprotein Metabolism in Hypertensive African-Americans
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4918; R01HL051536 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hyperinsulinism; Hypertension; Insulin Resistance
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hyperinsulinism; Hypertension; Insulin Resistance

SUMMARY:
To study relationships among lipoprotein metabolism, hypertension, and hyperinsulinemia-insulin resistance in African American males and females. The study was part of a Collaborative Project on Minority Health which investigated the mechanisms by which insulin contributes to cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of the initiative "Collaborative Projects (R01s) on Minority Health". The concept for the initiative was developed by the NHLBI staff after the 1993 Report of the Committee on Appropriations, House of Representatives, encouraged the NHLBI to establish minority centers to facilitate the diagnosis and treatment of cardiovascular diseases. The initiative was approved at the September 1992 National Heart, Lung, and Blood Advisory Council and released in October 1992.

Julian Marsh was one of three investigators in a collaborative program with Bonita Falkner as Program Coordinator.

DESIGN NARRATIVE:

In a sub-set of subjects with either high or low plasma insulin levels after a glucose challenge (insulin sensitive or insulin resistant), the investigators determined the fractional and absolute synthesis and catabolic rates of apolipoproteins B and A-I, the dominant lipoproteins of Low Density Lipoprotein (LDL) and High Density Lipoprotein (HDL). They used stable isotopes and multicompartmental kinetic analysis following an oral bolus dose of deuteroleucine. They hypothesized that in hypertensive African Americans with hyperinsulinemia, more of the smaller Very Low Density (VLDL) particles are secreted and converted to LDL.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1998-08 (Actual)

REFERENCES:
- [Background] Sumner AE, Kushner H, Tulenko TN, Falkner B, Marsh JB. The relationship in African-Americans of sex differences in insulin-mediated suppression of nonesterified fatty acids to sex differences in fasting triglyceride levels. Metabolism. 1997 Apr;46(4):400-5. doi: 10.1016/s0026-0495(97)90055-x. PMID 9109843
- [Background] Sumner AE, Kushner H, Lakota CA, Falkner B, Marsh JB. Gender differences in insulin-induced free fatty acid suppression: studies in an African American population. Lipids. 1996 Mar;31 Suppl:S275-8. doi: 10.1007/BF02637090. PMID 8729133
- [Background] Sumner AE, Falkner B, Diffenderfer MR, Barrett PH, Marsh JB. A study of the metabolism of apolipoprotein B100 in relation to insulin resistance in African American males. Proc Soc Exp Biol Med. 1999 Sep;221(4):352-60. doi: 10.1046/j.1525-1373.1999.d01-92.x. PMID 10460697